CLINICAL TRIAL: NCT03257566
Title: Risk Factors of Incidence of Hypothyroidism in Patients With Type 1 Diabetes
Brief Title: Hypothyroidism in Patients With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Romany Safwat, principal investigator, Assiut University
Other Study IDs: rfihtptd
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Therefore, for early detection of hypothyroidism in children with type 1 diabetes, it is suggested to measure anti-thyroid antibodies and thyroid stimulating hormone at disease onset and in yearly intervals after the age of 12 yr. Furthermore, the International Society for Pediatric and Adolescent Diabetes Consensus Clinical Guidelines recommend the screening of thyroid function by analysing circulating thyroid stimulating hormone at the diagnosis of diabetes and, thereafter every 2nd yr. in asymptomatic individuals without goitre and more frequent if goitre present .

DETAILED DESCRIPTION:
Type 1 diabetes is an organ-specific autoimmune disease characterized by the selective destruction of pancreatic β-cells. The histopathology of type 1 diabetes is defined by a decreased β-cell mass infiltration of mononuclear cells into the islets of Langerhans , this lesion was later called 'insulitis', and it is the hallmark of the disease .

Insulitis was observed in 70% of patients with acute onset type 1 diabetes and concluded that this disease was caused by a β-cell-specific autoimmune process .

Furthermore, in a study demonstrated cellular autoimmunity in patients with type 1 diabetes using the leukocyte migration test and speculated that cellular hypersensitivity was the counter part of lymphocytic infiltration in islets . Therefore, it is speculated that cell-mediated immunity could play an important part in the pathogenesis of type 1 diabetes .

As a view suggesting that type 1 diabetes is an autoimmune disease, there is some evidence that type 1 diabetes is often complicated with other autoimmune diseases or that anti-islet antibodies precede the clinical onset of the disease.

So, it is found that type 1 diabetes is frequently associated with other organ-specific autoimmune diseases, including hypothyroidism , pernicious anaemia, and idiopathic Addison's disease .The most common coexisting organ autoimmune disease is hypothyroidism (>90%), the prevalence of anti-thyroid autoantibodies in children with type 1 diabetes at disease onset is about 20% .

It is generally accepted that is a T cell-mediated autoimmune disease and that circulating autoantibodies to various islet cell antigens are induced following the destruction of pancreatic β cells .

Furthermore, it is reported that the prevalence of anti-thyroid antibodies increases with increasing age and that the presence of anti-thyroid antibodies at diagnosis of type 1 diabetes predicts the development of future thyroid disease as patients with antithyroid antibodies are 18 times more likely to develop thyroid disease than patients without anti-thyroid antibodies .

Therefore, for early detection of hypothyroidism in children with type 1 diabetes, it is suggested to measure anti-thyroid antibodies and thyroid stimulating hormone at disease onset and in yearly intervals after the age of 12 yr. Furthermore, the International Society for Pediatric and Adolescent Diabetes Consensus Clinical Guidelines recommend the screening of thyroid function by analysing circulating thyroid stimulating hormone at the diagnosis of diabetes and, thereafter every 2nd yr. in asymptomatic individuals without goitre and more frequent if goitre present .

ELIGIBILITY:
Inclusion Criteria:

- Children with type 1 diabetes aging between 8 - 15 y .

Exclusion Criteria:

1. Cases with hyperthyroidism .
2. Areas known to have endemic goitre due to nutritional iodine deficiency .
3. History of maternal hypothyroidism and / or congenital hypothyroidism .
4. Children known to be normoglycaemic with already presented thyroid dysfunction .
5. Children with multiple endocrinopathies .
6. Children under treatment with drugs inducing hypothyroidism like amiodarone , lithium .
7. Children under treatment with drugs affecting insulin secretion like steroids , growth hormone therapy .

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be applied on children with type 1 diabetes attending Diabetes Clinic at Sidy Galal Health Assurance Clinic in Assuit , aging between 8 - 15 yrs .
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Screening the incidence of hypothyroidism in patients with type 1 diabetes | after 1-2 years after diagnosis of Diabetes
  Measuring of thyroid stimulating hormone in patients with type 1 diabetes

IPD SHARING:
Plan to Share IPD: Undecided